CLINICAL TRIAL: NCT03687801
Title: Clinically Implementing Online Hearing Support
Brief Title: Clinically Implementing Online Hearing Support Within Hearing Organization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sodra Alvsborgs Hospital (Other)
Responsible Party: Principal Investigator, Milijana Malmberg, Principal Investigator, Sodra Alvsborgs Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: e-Hearing
Record Dates: First submitted 2018-09-20; First posted 2018-09-27 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Hearing Impairment
Keywords: audiologic rehabilitation; hearing loss; patient education; patient participation; structured rehabilitation; internet interventions; counseling
MeSH Terms: conditions — Hearing Loss; Patient Participation | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online hearing support (Experimental): The intervention group will have access to online hearing support for five weeks. The online hearing support will include a program that consists of three elements: 1) reading material; 2) reading instructions and weekly assignments related to the reading material; and 3) online and telephone interaction with a professional.
  Interventions: Behavioral: Online hearing support
- Standard care (Active Comparator): The control group will have access to traditional support that the Hearing Organization provides ("standard care").
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Online hearing support — The intervention group will follow an online hearing support for five weeks
  Arms: Online hearing support
Behavioral: Standard care — The control group will follow standard care during the time the intervention group receives online haring support
  Arms: Standard care

SUMMARY:
Previous research has proposed employing telehealth in hearing healthcare to improve clinical care and increase access to hearing services. Several studies have shown that hearing support can be carried out without in-person meetings and lead to significant benefits for hearing aid users. Interventions for persons with hearing impairment improve communication and improve outcomes more than hearing aid use alone.

The first purpose of this study is needs-oriented and the second purpose is research-oriented. The needs-oriented purpose of this project is to, via a national website of health information and services for Sweden, provide needed online support to hearing aid users. The research-oriented purpose of this project is to document the effectiveness of the online support compared to traditional support that the Hearing Organization, provides ("standard care").

DETAILED DESCRIPTION:
Aural rehabilitation The most common approach to hearing impairment is hearing aid fitting as a part of aural rehabilitation (AR). In Sweden, approximately 50% of those who could benefit from hearing aids are fitted with them, and nearly half of those use their hearing aids to a considerable extent every day. Despite addressing the hearing impairment with hearing aids, many hearing aid users experience substantial communication difficulties that can affect their performance in daily life situations. This could cause patients to stop using their hearing aids, which may negatively affect their interpersonal interactions and involvement in community life.

Adjusting to hearing impairment involves more than just hearing aid fitting, although hearing aid fitting is a step in the right direction. Additional steps within AR, such as learning about the condition and providing perceptual training and counseling, need to be included in order to minimize the negative effects of a hearing impairment on social interactions and quality of life. These additional steps can effectively be included variously throughout the AR (separately or in combination, and individually or in groups), they may increase hearing aid use and satisfaction, and can be performed as an adjunct to or a supplement for hearing aid fitting. However, even though combining these additional steps with hearing aid use has proven to be beneficial, most hearing aid users are unaware of and are not offered any other rehabilitation measures than hearing aid fitting. This deficiency could be due to clinicians experiencing lack of time and difficulties scheduling interventions in addition to hearing aid fitting. It could also be due to the presumably increased costs of adding extra support to hearing aid fitting. These aspects could hinder audiologist's in general clinical practice from providing holistic care. Thus, the overall availability of comprehensive AR is low.

Internet interventions Online interventions and healthcare information is cost-effective. Online hearing healthcare has increased in recent years and is empowering for persons with hearing impairment. Telehealth (i.e., telephone and internet) offers a more cost-effective approach to hearing healthcare and increases the possibilities for the audiologist to reach out to persons with hearing impairment. Previous research has proposed employing telehealth in hearing healthcare to improve clinical care and increase access to hearing services.

Effective internet interventions have four important interactive design features: 1) social context and support, 2) contacts with intervention, 3) tailoring, and 4) self-management. Patient participation is central for self-management to be successful. For example, a person with hearing impairment can apply knowledge obtained in communication training to reduce hearing-related problems. The role of the audiologist in delivering social contact and support, and contacts with the intervention, seems to be of particular importance in online audiology interventions.

Purpose With this project we want to provide online support to hearing aid users. Further on, we want to document the effectiveness of the online support compared to traditional support that the Hearing Organization, VGR, provides ("standard care").

The needs-oriented purpose: The project is a part of a collaboration between 1177 Care-Guide and region Vastra Gotaland (VGR). 1177 Care-Guide is a national website of health information and services for Sweden. Every region customizes its 1177 Care-Guide. Regions use the 1177 Care-Guide platform to provide online services. The needs-oriented purpose of this project is to, via 1177, provide needed online support to hearing aid users. The research-oriented purpose of this project is to document the effectiveness of the online support compared to traditional support that the Hearing Organization, VGR, provides ("standard care"). Traditional support ("standard care") in Sweden differs across and within counties, in particular in terms of the number of visits and the content of comprehensive AR. The costs of amplification for the person with hearing impairment may also vary across counties.

ELIGIBILITY:
Inclusion Criteria:

* the hearing aid users to be 20 yr of age or above,
* the hearing aid users to have completed a hearing aid fitting at least 3 months before the study began (regardless of hearing aid manufacturer, model, or hearing aid outcomes),
* the hearing aid users to have a Hearing Handicap Inventory for the Elderly (HHIE) score of >20 points (indicative of some residual self-reported hearing problems).

Exclusion Criteria:

* the hearing aid users who are not fulfilling the conditions to participate.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Change is assessed for the Hearing Handicap Inventory for the Elderly (HHIE) | change from baseline HHIE at 5 weeks, change from baseline HHIE at 6 months, change from baseline HHIE at 1 year
  The HHIE measures the experience of hearing loss in older people by focusing on the psychosocial and emotional effects of hearing loss. Higher score reflects a higher self-reported hearing problem. Minimum score for the total scale (reported) is 0 and maximum score is 100 points.

SECONDARY OUTCOMES:
Change is assessed for the Communication Strategies Scale (CSS) | change from baseline CSS at 5 weeks, change from baseline CSS at 6 months, change from baseline CSS at 1 year
  CSS (from the Communication Profile for the Hearing Impaired) The CSS is designed to analyze participants' behavior in various communication situations via three subscales: maladaptive behaviors (9 questions that analyze behaviors that hinder communication) and verbal strategies and nonverbal strategies (16 items related to strategies that can enhance communication). The 1 to 5 scoring reflects how frequently a specific situation or behavior occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Milijana Malmberg, PhD, Principal Investigator — Hörselverksamheten, Habilitering & Hälsa
Locations (1):
- Hearing Clinic, Hearing Organization, Borås, Vastra Gotalandsregion, Sweden

IPD SHARING:
Plan to Share IPD: No